CLINICAL TRIAL: NCT07176013
Title: Immediate and Cumulative Effects of Meditation on Voice Therapy Using Immersive Virtual Reality (IVR)
Brief Title: Immersive Virtual Reality Meditation in Voice Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Bradley Hoff, Speech-Language Pathologist, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-24-01217
Record Dates: First submitted 2025-07-30; First posted 2025-09-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Voice Disorders
Keywords: Virtual Reality; Immersive; Mindfulness; Meditation; Voice
MeSH Terms: conditions — Voice Disorders | interventions — Meditation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Meditation with VR (Experimental): Those who receive meditation in immersive virtual reality prior to voice therapy each of the 4 sessions.
  Interventions: Behavioral: Voice therapy; Behavioral: Meditation; Device: Virtual Reality
- Meditation without VR (Experimental): Those who receive meditation with verbal guidance only prior to voice therapy each of the 4 sessions.
  Interventions: Behavioral: Voice therapy; Behavioral: Meditation
- No Meditation (Sham Comparator): Those who receive standard voice therapy with no meditation.
  Interventions: Behavioral: Voice therapy

INTERVENTIONS:
Behavioral: Voice therapy — All patients will receive a course of voice therapy as normal.
Behavioral: Meditation — Meditation at the start of each session. (each session is 30 minutes)
  Arms: Meditation with VR; Meditation without VR
Device: Virtual Reality — TRIPP application in the Meta Quest 2 Virtual Reality Headset.
  Arms: Meditation with VR

SUMMARY:
This study aims to explore the feasibility of incorporating regular guided meditations via immersive virtual reality (IVR) at the start of voice therapy sessions to facilitate better learning and retention of treatment. The study will involve 30 participants, and use the TRIPP application with the Meta Quest 2 virtual reality headset, known for its immersive meditation experiences designed to calm or focus the user. The objective is to investigate the immediate effects of meditation/mindfulness in IVR on vocal production, with the goal of improving self-regulation, attentional focus, and reducing vocal hyperfunction. IVR has been utilized in mental health settings and exposure therapy for various conditions, but its application in voice therapy, particularly for anxiety reduction through fully immersive meditation, remains unexplored. The study seeks to determine whether IVR can enhance therapy outcomes by improving engagement, attention, and vocal control in individuals undergoing voice therapy, potentially maximizing treatment gains. Through this research, the aim is to assess the efficacy of IVR in enhancing voice therapy interventions and addressing the unique challenges posed by stress and anxiety in voice users.

ELIGIBILITY:
Inclusion Criteria:

* Patients with voice disorders, difficulties or laryngeal hypersensitivity, and who also have anxiety
* Must have availability to participate for entire course of 5 consistent weeks

Exclusion Criteria:

* Anyone not meeting inclusion criteria
* Presence of any additional medical condition significantly affecting:

  * Respiratory function (e.g., advanced lung disease)
  * Laryngeal function (e.g., status-post deep brain stimulation)
  * Lingual function
  * Velopharyngeal function (e.g., laryngectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Phonation Time (MPT) | at each therapy session (approximately 1 week apart over 4 weeks)
  MPT will be used to assess participants' maximum phonation time. The speech evaluator instructs the patient to take a comfortable breath and then produce the sound /a/ for as long as possible. The task is performed twice, and the maximum duration of the two measurements is used.
Noise-to-Harmonic Ratio (NHR) | Pre-intervention (within 1 week before first session) and post-intervention (within 1 week after final session
  NHR is a parameter in MDVP that represents ratio of non-harmonic and harmonic waves in a certain sound wave period. NHR describes the quality of the amount of noise in the sound. Inadequate closure of the vocal cords and periodic vibrations of the vocal cords cause excessive air flow as it passes through the vocal cords, causing turbulence and noise. Normal and periodic sound signals will have a small NHR, while dysphonia sound signals will have a large NHR value.
Cepstral Peak Prominence (CPPS) | Pre-intervention (within 1 week before first session) and post-intervention (within 1 week after final session
  Cepstral Peak Prominence (CPPS) is an indicator of voice quality. It is measured in decibels. An increase in CPPS value indicates an improvement in voice symptoms.
Acoustic Vocal Quality Index (AVQI) | Pre-intervention (within 1 week before first session) and post-intervention (within 1 week after final session
  The acoustic voice quality index (AVQI) is a multiparametric score to quantify vocal quality. It is based on a weighted combination of 6 voice parameters: smoothed cepstral peak prominence (CPPS), harmonics-to-noise ratio (HNR), shimmer local (SL), shimmer local dB (SLdB), general slope of the spectrum (slope) and tilt of the regression line through the spectrum (tilt). The formula is constructed as 9.072 - 0.245 × CPPs - 0.161 × HNR - 0.470 × SL + 6.158 × SLdB - 0.071 × Slope - 0.170 × Tilt and ranges from 0 to 10. A lower score correlates with a better vocal quality.

SECONDARY OUTCOMES:
Voice Handicap Index | Pre-intervention (within 1 week before first session) and post-intervention (within 1 week after final session
  The Voice Handicap Index (VHI) is a validated 10-item questionnaire measuring the impact of voice challenges on quality of life (QOL). Scores range from 0 to 40, with higher scores indicating greater perceived voice handicap and negative impact on daily functioning.
State Trait Anxiety Inventory Y-1 (STAI-1), long form | Pre-intervention (within 1 week before first session) and post-intervention (within 1 week after final session
  The State Anxiety Inventory (STAI Y-1) long form assess the severity of current state of anxiety in the moment, with a minimum score of 40 and max of 80, where scores >37 indicates moderate-severe state anxiety. Higher score indicates more severity of anxiety
State Trait Anxiety Inventory Y-1 (STAY Y-1), short form | Immediately pre- and immediately post-meditation in each therapy session, over approximately 4 weeks
  The State Anxiety Inventory-Short Form (STAI Y-1) assesses severity of current state of anxiety in the moment to determine immediate effects of meditation. Scores range from 20-40. Higher score indicates more severity of anxiety.
State Trait Anxiety Inventory Y-2 (STAI Y-2), long form | Pre-intervention (within 1 week before first session) and post-intervention (within 1 week after final session
  The State Trait Anxiety Inventory (STAI Y-2) assesses severity of anxiety relative to how the patient "generally" feels. Scores range 40-80, with scores >37 indicating moderate-severe trait anxiety. Higher score indicates more severity of anxiety.
Vocal Fatigue Index | Pre-intervention (within 1 week before first session) and post-intervention (within 1 week after final session
  The Vocal Fatigue Index (VFI) is a validated questionnaire designed to measure three distinct dimensions of vocal fatigue and voice disorders. It evaluates scores across three subscales:
  Fatigue and Avoidance (Part 1): Scores range from 0 to 44, with scores ≥24 indicating severity.
  Physical Discomfort (Part 2): Scores range from 0 to 20, with scores ≥7 indicating severity.
  Improvement with Rest (Part 3): Scores range from 0 to 12, with scores ≤7 indicating severity.
  Higher scores on Parts 1 and 2, and lower scores on Part 3, indicate greater voice disorder severity. The VFI is intended to be used for the score of each subscale individually and is not validated to measure severity based on the composite score. However, the maximum total score across all three subscales is 79.
CAPE-V, Consensus on Auditory-Perceptual Evaluation of Voice | Pre-intervention (within 1 week before first session) and post-intervention (within 1 week after final session
  A subjective auditory-perceptual evaluation to judge the severity of dysphonia from the standpoint of expert clinician raters (at least 2 for each sample, not including the treating clinician). Scale of severity overall from 0-100. Higher score indicates more severity of symptoms.
Heart rate measured in beats per minute | Immediately pre- and immediately post-meditation in each therapy session, over approximately 4 weeks
  Heart rate (HR) is measured in beats per minute (bpm) using a standard hospital-provided pulse oximeter to assess cardiovascular function.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley R Hoff, MA, CCC-SLP, Principal Investigator — Icahn School of Medicine at Mount Sinai, Department of Otolaryngology; Ümit Daşdöğen, Ph.D., CCC-SLP, Study Director — Icahn School of Medicine at Mount Sinai, Department of Otolaryngology
Locations (1):
- Mount Sinai Downtown Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. Any purpose. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be determined).